CLINICAL TRIAL: NCT00472368
Title: An Open-label, Single Center, Study to Determine the Absorption, Distribution, Metabolism, and Excretion (ADME) of LBH589 After a Single Oral Administration of 20 mg (14C) LBH589 in Advanced Cancer Patients
Brief Title: A Study to Determine the Absorption, Distribution, Metabolism, and Excretion of LBH589
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2108
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Cancer Patients With Advanced Solid Tumors Including Lymphoma or Chronic Hematological Malignancies
Keywords: Advanced cancer; lymphoma; chronic hematological malignancies; adult
MeSH Terms: conditions — Lymphoma | interventions — Panobinostat

ARMS (1):
- LBH589 (Experimental)
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589
  Other Names: Panobinostat

SUMMARY:
This single center study will help determine the absorption, metabolism, and excretion of LBH589 and to assess the safety and efficacy of LBH589 in advanced cancer patients for whom no standard therapy exists.

ELIGIBILITY:
Inclusion criteria

* Histologically or cytologically confirmed cancer patients including solid tumors, lymphoma, or chronic hematological malignancies with progression on prior standard therapies.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of < 2
* Normal renal and hepatic function

Exclusion criteria

* Patients with central nervous system (CNS) involvement or brain metastases
* Patients who have received chemotherapy, any investigational drug, undergone major surgery, or received wide field radiotherapy less than 4 weeks ago
* Patients with congenital long QT syndrome or uncontrolled hypertension
* Patients with a myocardial infarction or unstable angina within 6 months
* Congestive heart failure
* Impairment of gastrointestinal (GI) function
* Use of any anti-cancer therapy
* Female patients who are pregnant or breast feeding

Other protocol inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Rates and routes of excretion of LBH589 and its metabolites in urine and feces following administration of a single oral dose of [14C] LBH589 | during the first 8 days on study
  oral dose of [14C] LBH589

SECONDARY OUTCOMES:
Safety Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Buffalo, New York, United States